CLINICAL TRIAL: NCT02399800
Title: Prospective Randomized Trial of EUS Guided Celiac Plexus Block for Chronic Pancreatitis
Brief Title: Celiac Plexus Block for Chronic Pancreatitis RCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, James Buxbaum, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-14-00134
Record Dates: First submitted 2015-01-11; First posted 2015-03-26 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Pancreatitis, Chronic; Pancreatitis
Keywords: pancreatitis, chronic; endosonography
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis | interventions — Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EUS with Celiac Block (Experimental): Celiac Block with triamcinolone and bupivicaine Intra Plexus Triamcinolone and Bupivicaine Injection
  Interventions: Procedure: Celiac Block with triamcinolone and bupivicaine; Drug: Intra Plexus Triamcinolone and Bupivicaine Injection
- EUS without Celiac Block (Active Comparator): Patients will undergo EUS but no celiac block will be performed
  Interventions: Procedure: No Celiac Block

INTERVENTIONS:
Procedure: Celiac Block with triamcinolone and bupivicaine — Endosonography of the pancreas performed following by analgesic injection
  Arms: EUS with Celiac Block
Procedure: No Celiac Block — EUS but no celiac block performed
  Arms: EUS without Celiac Block
Drug: Intra Plexus Triamcinolone and Bupivicaine Injection — Injection of Triamcinolone and Bupivicaine into celiac plexus for pain relief
  Other Names: kenalog
  Arms: EUS with Celiac Block

SUMMARY:
Rationale: Chronic pancreatitis is a chronic inflammatory disease of the pancreas which results in debilitating abdominal pain, decreased productivity and increased health care costs. Endoscopic ultrasound (EUS) guided celiac plexus block (CPB) is routinely used to treat pain related to chronic pancreatitis. While EUS guided neurolysis for pancreatic cancer has significant efficacy, the benefit of CPB for chronic pancreatitis pain is controversial and has not been studied in a rigorous manner.

Objective: To assess whether EUS guided celiac plexus block decreases suffering, hospitalization, and opiate requirements related to chronic pancreatitis pain.

Population: Patients undergoing EUS at Los Angeles County Hospital for painful chronic pancreatitis.

Methods: Patients undergoing EUS to evaluate chronic pancreatitis with a typical visual analogue pain score >3, regular opiate use, and M ANNHEIM chronic pancreatitis score >6 will be eligible.

Study Arms: Patients will be randomized to 1) diagnostic endoscopic ultrasound 2) endoscopic ultrasound with celiac plexus block

Study Outcomes: The primary outcome will be a decrease in chronic pancreatitis pain assessed by the visual analogue scale and M ANNHEIM system at 24 weeks compared to immediately prior to the block. The ability to work and conduct normal activities, opiate medication requirements, and a Careprep symptom assessment at 24 weeks will also be compared prior to the block.

Analytic Plan: The projected response rate to EUS guided CPB is 52%. Given known 30% placebo response in patients with pain related to chronic pancreatitis we anticipate that 83 patients will need to participate to demonstrate a difference. We aim to enroll 90 patients in this study.

DETAILED DESCRIPTION:
1.0 Background and Hypothesis: Chronic pancreatitis is an inflammatory disease of the pancreas characterized by painful scarring and loss of glandular function.The prevalence of chronic pancreatitis in the United States is estimated to be 0.2 to 5% and results in 86,000 hospitalizations. The majority of patients with chronic pancreatitis will develop significant abdominal pain which is debilitating and results in a significant burden on the health care system.

Multiple approaches, including pancreatic enzymes, narcotic analgesia, celiac plexus block and surgical ganglionectomy have been used to treat pancreatic pain with variable success. Injection of local anesthesia agents and steroids into the celiac plexus for pain control has been used for many years via both surgical and percutaneous approaches. Topical therapy theoretically prevents the conduction of painful stimuli from the pancreas and addresses inflammatory changes in the afferent nerves themselves. Splanchnic nerves pass from the pancreas to the thoracic root ganglia via the celiac ganglia which are the target for intervention. Nerve changes in chronic pancreatitis including perineural inflammation, altered diameter, and upregulation of pain neuropeptides (including Substance P) are associated with increased sensitivity to stimuli from the pancreas (distension and inflammation) as well as pain independent of stimuli (neuropathic). Endoscopic ultrasound allows for close proximity, high resolution assessment of the gastrointestinal tract wall and adjacent anatomic structures. Physicians are able to perform EUS-guided celiac plexus injections in the outpatient setting under conscious sedation. The EUS guided approach offers better visualization of the celiac region and direct access to the celiac plexus. EUS guided celiac plexus block is a core part of the routine care of patients at Los Angeles County Hospital with chronic pancreatitis. Celiac plexus block is a recommendation for refractory chronic pancreatitis pain by the European Society of Gastrointestinal Endoscopy (ESGE).

Several studies have shown that EUS-guided CPB has a beneficial role in treating pain caused by chronic pancreatitis. A randomized trial by Gress et al looked at the efficacy of EUS-guided versus CT-guided celiac plexus block for controlling abdominal pain of chronic pancreatitis in 18 patients. They found significant improvement in pain symptoms in patients randomized to EUS-guided celiac plexus block over a mean time period of 10 weeks. A study by the same group showed an improvement in overall pain score in 55% at 4 and 8 weeks of follow-up in 90 patients. Adverse events including diarrhea and infection occurred in 3%. A comprehensive review by Kaufman et al in 2010 evaluated the efficacy of EUS-guided celiac plexus block and celiac plexus neurolysis in alleviating chronic abdominal pain due to chronic pancreatitis and pancreatic cancer respectively. A total of 6 studies were included in their analysis, comprising 221 patients, and found that EUS-guided celiac plexus block was effective in 51.46% of patients with chronic pancreatitis. EUS-guided celiac plexus neurolysis (with alcohol) was effective in 72.54% of those with pancreas cancer.

These modest improvement for celiac block for chronic pancreatitis (especially in comparison to celiac plexus neurolysis in pancreas cancer) have led some investigators to question whether EUS guided celiac plexus block is an effective treatment for chronic pancreatitis pain despite its routine use. Prospective randomized controlled studies examining the efficacy of endoscopic ultrasound guided celiac plexus block are lacking.

2.0 Objectives and Purpose Our aim is to perform a pilot randomized trial to gauge the degree to which celiac plexus block performed under endoscopic ultrasound guidance will benefit patients with chronic pancreatitis. We will assess whether celiac plexus block significantly decreases pain scores, hospitalization, and pain medication requirements and increases the ability to return to normal activities.

3.0 Study Design Patients presenting to the Los Angeles County Medical Center and Gastroenterology Clinic with chronic upper abdominal pain are the focus population of this study. Patients who are undergoing endoscopic ultrasound for standard clinical care to assess for chronic pancreatitis will be enrolled. They must have a M-ANNHEIM severity score of 6 or greater. Additionally, they must have at least intermittent if not chronic pain of intensity >3 on the visual analogue scale requiring opiate medication.

The procedures will be performed by experienced endosonographers. The EUS-guided celiac plexus block will be performed under the guidance of linear array endosonography. A visual exam will first be performed with the EUS scope or a standard endoscope. Patients found to have a significant peptic ulcer or other mucosal abnormality will be excluded as the symptoms may be secondary to peptic disease. An EUS exam will then be performed to determine whether the patient has findings of chronic pancreatitis. The diagnosis of chronic pancreatitis will be confirmed based on EUS criteria (meeting four or more criteria of hyperechoic foci, hyperechoic strands, lobularity, cysts, stones, dilation of the main pancreatic duct, irregular pancreatic-duct margins, presence of side branches and hyperechoic pancreatic duct-margins).

Those who are confirmed to have chronic pancreatitis will be randomized (1:1) during the procedure to celiac plexus block versus no injection treatment. Randomization will be performed using a computer program with concealed allocation. The research coordinator obtaining data for follow up visits and the patient will be blinded to randomization. The endosonographer will not be blinded. Ninety patients will be enrolled (see statistical considerations for sample size calculation).

Those randomized to control will undergo EUS and confirmation of chronic pancreatitis but not celiac plexus block. Patients in the treatment group will receive celiac plexus block with 10mL 0.25% bupivacaine and 2ml (40mg/cc) triamcinolone which are the standard doses. The 22 gauge needle will be inserted into the base of the celiac plexus via the transgastric approach and a single injection will be performed. An intravenous antibiotic will be administered at the time of the block to those in the celiac plexus block group with the specific agent depending on the patient's allergy profile. The research coordinator obtaining data for follow up visits and the patient will be blinded to the details of the block (or lack thereof) procedure but it will be recorded.

Following the procedure standard recovery room monitoring including assessment of blood pressure be performed for 2 hours for both groups. Periprocedural fluid and antibiotic use for celiac plexus block is not standardized and will be at the discretion of the endoscopist performing the cases.

Patients will be assessed before the procedure, immediately afterward, and at 2 weeks, 6 weeks, 3 months, and 6 months following the procedure. At the initial assessment and follow up visits Visual analogue pain scores will be recorded as well as an assessment of the ability to work and conduct activities of daily living. Pain medication requirements and whether symptoms are alleviated by analgesic or disrupt sleep will be noted. The M-ANNHEIM scoring system will be used to gauge symptoms as well.

Additionally, patients will complete a focused version of the online CarePrep Program during each visit. The Online CarePrep (OCA) program is used to clinically evaluate patients with complex symptoms or conditions generally characterized significant physical symptoms, psychosocial issues, impaired quality-of-life and functional status, disability, and substance abuse. It has an online format that has been successfully used by outpatient with various gastrointestinal illness to report multifactorial symptoms. When performed prior to appointments it appears to facilitate efficient and productive medical visits.

4.1 Side effects/Toxicities to be monitored:

4.11 Three most common complications from celiac plexus block include hypotension, transient diarrhea, transient increase in pain. Extraordinarily rare/theoretical complications include paralysis, pneumothorax, loss of sphincter function, retroperitoneal bleeding, renal puncture and prolonged gastroparesis.

4.12 Long term toxicities to be monitored after completion of the celiac block during the 6 months the patients are followed.

4.2 Dosage changed based on toxicity There will be no dosage adjustments as the procedure will be performed once during the study period.

4.3 Adverse Event Reporting: 4.31 Type of event to be reported and timing of reports. If patients develop adverse events including hypotension, transient diarrhea, transient increase in pain, or less common complications of unilateral paresis or paraplegia, pneumothorax, loss of sphincter function, retroperitoneal bleeding, renal puncture, prolonged gastroparesis or infection, this will be reported to the principal investigators and will be reviewed by the study team as well as two staff physicians in the gastroenterology division who are not part of the study team. This will also be reported to the IRB.

If patients experience any further events that are detected during follow up these will be coded as A) related to study or B) not related to study. Their severity and A) whether they were expected or B) not expected will also be recorded. These complications will also be reported to the principal investigators and will be reviewed by the study team as well as two staff physicians in the gastroenterology division who are not party of the study team. They will also be reported to the IRB.

4.32 Places for submitting reports: Adverse events will be reported to the IRB and data safety monitoring committee.

4.4 Data Monitoring Committee: The data safety monitoring committee will include the principal investigators from medicine/gastroenterology as well as the entire study team. Two outside senior physician from gastroenterology or surgery will also be asked to participate. Meetings will be convened if adverse events potentially related to the celiac block occur.

5.0 Statistical Considerations Descriptive statistics will be performed for each group, and comparisons made to determine if the groups are balanced on the stratification factor of type of pancreatitis. Patient characteristics will be compared between groups as well to determine if there is imbalance of other possible covariates. We expect that there will be patients with chronic pancreatitis secondary to congenital abnormalities of the pancreatic duct, ethanol abuse, familial, and idiopathic etiologies.

The sample size of 90 patients was chosen based on preliminary sample size calculations. Based on recent studies 30% of patients with pancreatitis type pain in the placebo arm will derive benefit.16 The predicted response rate of 51.5% for EUS guided celiac block was based on the large review by Kaufmann et al. For a 2 sided alpha of 0.05 and a power of 0.80, 83 patients would be necessary to show a difference. Statistical analyses will be performed by biostatisticians at the Biostatistical and Bioinformatics Resource Group within the SC CTSI.

ELIGIBILITY:
Inclusion Criteria:

* Presentation with upper abdominal pain suggestive of pancreatitis who are undergoing EUS for evaluation
* M ANNHEIM severity index of 6 or greater to be included
* Intermittent episodes of pain>3 requiring opiate medication

Exclusion Criteria:

* Patients who have allergic reactions to steroids or bupivacaine
* INR >1.6
* platelets <75
* decompensated cirrhosis
* incarcerated
* <18 years old
* unable to give informed consent
* peptic ulcer disease
* ongoing substance or alcohol use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-12; Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
Long Term CHANGE in Pain Scores | 24 weeks
  Primary outcomes will be the CHANGE pain score (as assessed by the visual-analogue-scale and M-ANNHEIM score assessed between time 0 and 24 weeks post procedure in those who undergo EUS without block (control) compared to those who undergo EUS with block

SECONDARY OUTCOMES:
Hospital re-admission | 24 weeks
  differences in number of hospital re-admissions for pancreatic pain assessed at 24 weeks between those who underwent the block and did not undergo the celiac block
CHANGE Pain medication requirements | 24 weeks
  CHANGE in pain medication requirement 24 weeks following celiac block in those who underwent EUS guided celiac block compared to those who did not
Procedure Complications | 2 weeks
  Post procedure complications include infection (defined as fever or increased WBC without an alternative cause), diarrhea (defined as 3 loose stools per day), or pancreatitis (defined as increased pain and lipase >3 X the upper limit of normal). Will be assessed 2 weeks after the procedure and compared between those who EUS with block compared to EUS without block

CONTACTS AND LOCATIONS:
Overall Officials: James Buxbaum, MD, Principal Investigator — Los Angels County Hospital
Locations (1):
- Los Angeles County Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sarles H. Etiopathogenesis and definition of chronic pancreatitis. Dig Dis Sci. 1986 Sep;31(9 Suppl):91S-107S. doi: 10.1007/BF01295992. PMID 3525051
- [Background] Wilcox CM. Tinkering with a tarnished technique: isn't it time to abandon celiac plexus blockade for the treatment of abdominal pain in chronic pancreatitis? Clin Gastroenterol Hepatol. 2012 Feb;10(2):106-8. doi: 10.1016/j.cgh.2011.10.039. Epub 2011 Nov 9. No abstract available. PMID 22079511
- [Background] Kozak LJ, Owings MF, Hall MJ. National Hospital Discharge Survey: 2002 annual summary with detailed diagnosis and procedure data. Vital Health Stat 13. 2005 Mar;(158):1-199. PMID 15853196
- [Background] Gress F, Schmitt C, Sherman S, Ciaccia D, Ikenberry S, Lehman G. Endoscopic ultrasound-guided celiac plexus block for managing abdominal pain associated with chronic pancreatitis: a prospective single center experience. Am J Gastroenterol. 2001 Feb;96(2):409-16. doi: 10.1111/j.1572-0241.2001.03551.x. PMID 11232683
- [Background] Drewes AM, Krarup AL, Detlefsen S, Malmstrom ML, Dimcevski G, Funch-Jensen P. Pain in chronic pancreatitis: the role of neuropathic pain mechanisms. Gut. 2008 Nov;57(11):1616-27. doi: 10.1136/gut.2007.146621. Epub 2008 Jun 19. PMID 18566105
- [Background] Goodman AJ, Gress FG. The endoscopic management of pain in chronic pancreatitis. Gastroenterol Res Pract. 2012;2012:860879. doi: 10.1155/2012/860879. Epub 2012 Mar 5. PMID 22550479
- [Background] Dumonceau JM, Delhaye M, Tringali A, Dominguez-Munoz JE, Poley JW, Arvanitaki M, Costamagna G, Costea F, Deviere J, Eisendrath P, Lakhtakia S, Reddy N, Fockens P, Ponchon T, Bruno M. Endoscopic treatment of chronic pancreatitis: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2012 Aug;44(8):784-800. doi: 10.1055/s-0032-1309840. Epub 2012 Jul 2. PMID 22752888
- [Background] Gress F, Schmitt C, Sherman S, Ikenberry S, Lehman G. A prospective randomized comparison of endoscopic ultrasound- and computed tomography-guided celiac plexus block for managing chronic pancreatitis pain. Am J Gastroenterol. 1999 Apr;94(4):900-5. doi: 10.1111/j.1572-0241.1999.01042.x. PMID 10201454
- [Background] Kaufman M, Singh G, Das S, Concha-Parra R, Erber J, Micames C, Gress F. Efficacy of endoscopic ultrasound-guided celiac plexus block and celiac plexus neurolysis for managing abdominal pain associated with chronic pancreatitis and pancreatic cancer. J Clin Gastroenterol. 2010 Feb;44(2):127-34. doi: 10.1097/MCG.0b013e3181bb854d. PMID 19826273
- [Background] Schneider A, Lohr JM, Singer MV. The M-ANNHEIM classification of chronic pancreatitis: introduction of a unifying classification system based on a review of previous classifications of the disease. J Gastroenterol. 2007 Feb;42(2):101-19. doi: 10.1007/s00535-006-1945-4. Epub 2007 Mar 12. PMID 17351799
- [Background] Varadarajulu S, Eltoum I, Tamhane A, Eloubeidi MA. Histopathologic correlates of noncalcific chronic pancreatitis by EUS: a prospective tissue characterization study. Gastrointest Endosc. 2007 Sep;66(3):501-9. doi: 10.1016/j.gie.2006.12.043. Epub 2007 Jul 20. PMID 17640639
- [Background] Kleykamp M. Unemployment, earnings and enrollment among post 9/11 veterans. Soc Sci Res. 2013 May;42(3):836-51. doi: 10.1016/j.ssresearch.2012.12.017. Epub 2013 Jan 7. PMID 23521998
- [Background] Eypasch E, Williams JI, Wood-Dauphinee S, Ure BM, Schmulling C, Neugebauer E, Troidl H. Gastrointestinal Quality of Life Index: development, validation and application of a new instrument. Br J Surg. 1995 Feb;82(2):216-22. doi: 10.1002/bjs.1800820229. PMID 7749697